CLINICAL TRIAL: NCT00072566
Title: Phase II Clinical Trial of Bevacizumab (NSC 704865) and Low Dose Oral Cyclophosphamide in Recurrent Ovarian Cancer, Primary Peritoneal Carcinoma
Brief Title: Bevacizumab and Low-Dose Cyclophosphamide in Treating Patients With Recurrent Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02562; NCI-2012-02562 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5789; CHNMC-PHII-45; CDR0000340522; CCC-PHII-45; PHII-45 (Other: City of Hope Comprehensive Cancer Center); 5789 (Other: CTEP); N01CM17101 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2012-12

CONDITIONS: Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma; Stage IV Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cyclophosphamide

ARMS (1):
- Treatment (bevacizumab, cyclophosphamide) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1, 8, and 15 for the first course and on days 1 and 15 for all subsequent courses. Patients also receive low-dose oral cyclophosphamide on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is to see if combining bevacizumab with low-dose cyclophosphamide works in treating patients with ovarian epithelial or primary peritoneal cancer that has come back or spread to other parts of the body. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining bevacizumab with cyclophosphamide may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the time to progression in patients with recurrent ovarian epithelial or primary peritoneal cancer treated with bevacizumab and low-dose cyclophosphamide.

Secondary I. Determine the response rate in patients treated with this regimen. II. Determine the toxicity of this regimen in these patients. III. Determine molecular correlates for response and outcomes in patients treated with this regimen.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on days 1, 8, and 15 for the first course and on days 1 and 15 for all subsequent courses. Patients also receive low-dose oral cyclophosphamide on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 23-55 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic ovarian epithelial or primary peritoneal cancer
* Unidimensionally measurable disease

  * Previously irradiated indicator lesions must have progressed after radiotherapy
* Received a platinum-containing regimen for primary disease
* No more than 2 prior chemotherapy regimens for recurrent disease

  * Must have received prior platinum-based chemotherapy for recurrent disease if it has been > 12 months since treatment for primary disease (except if hypersensitivity to platinum has developed)
  * Rechallenge with the same platinum-based regimen is considered 1 prior regimen
* No history or clinical evidence of CNS disease, including primary brain tumor
* No brain metastases
* Performance status - SWOG 0-2
* At least 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding diathesis
* No coagulopathy
* Bilirubin no greater than 1.5 times normal
* ALT or AST no greater than 3 times upper limit of normal
* INR less than 1.5 (for patients receiving warfarin)
* Creatinine no greater than 1.5 times normal
* No proteinuria (less than 1+)
* Proteinuria less than 500 mg/24-hour urine collection
* No prior deep vein thrombosis
* No prior stroke
* No clinically significant cardiovascular disease
* None of the following within the past year:

  * Uncontrolled hypertension
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Grade II or greater peripheral vascular disease
* None of the following within the past 6 months:

  * Unstable angina
  * Myocardial infarction
  * Transient ischemic attack
  * Cerebrovascular accident
  * Other arterial thromboembolic event
* No clinically significant peripheral artery disease
* No active infection requiring parenteral antibiotics
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No serious, non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 28 days
* No seizures not controlled with standard medical therapy
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * All prior invasive malignancies must be in complete remission
* No other concurrent medical, psychological, or social condition that would preclude study participation
* No prior antiangiogenesis agents
* See Disease Characteristics
* Recovered from prior chemotherapy
* See Disease Characteristics
* Recovered from prior radiotherapy
* More than 28 days since prior major surgical procedure or open biopsy and recovered
* At least 3 weeks since prior therapy directed at the malignancy
* No recent or concurrent full-dose anticoagulants or thrombolytic agents

  * Anticoagulants to maintain patency of preexisting, permanent indwelling IV catheters allowed
* No concurrent chronic daily aspirin (greater than 325 mg/day) or nonsteroidal anti-inflammatory drugs known to inhibit platelet function

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Bevacizumab, Cyclophosphamide): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1, 8, and 15 for the first course and on days 1 and 15 for all subsequent courses. Patients also receive low-dose oral cyclophosphamide 50 mg/d on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  bevacizumab: Given IV
  cyclophosphamide: Given PO
Period: Overall Study
Arm/Group | Treatment (Bevacizumab, Cyclophosphamide)
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 60 [31 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression
Description: Time from treatment initiation to disease progresion calculated using the method of Kaplan-Meier. RECIST v1.0 was used to evaluate response. Progression was defined as a 20% or greater increase in the sums of the longest dimensions of target lesions, or the appearance of new lesions within 8 weeks of study entry.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 70
months | 7.2 [5.3 to 8.7]

2. Secondary Outcome: Response Rate Based on the RECIST
Description: Percentage of patients with a confirmed partial or complete response using RECIST v1.0 criteria. Complete response was defined as the disapperance of all target and nontarget lesions, no evidence of new lesions and normalization of CA-125; Partial response was defined as a 30% or greater reduction in the sum of the longest dimensions of all target lesions and no unequivocal progression of nontarget lesions, lasting at least 4 weeks.
Time Frame: Up to 3 years
Measure: Number; unit: percentage of responding patients
Arm/Group | Treatment (Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 70
percentage of responding patients | 24

3. Secondary Outcome: Median Overall Survival
Description: Calculated using the method of Kaplan-Meier.
Time Frame: Time from first day of treatment to time of death due to any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 70
months | 16.9 [11.4 to 25.2]

ADVERSE EVENTS:
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Bevacizumab, Cyclophosphamide)
Serious Adverse Events (participants affected / at risk) | 23/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab, Cyclophosphamide) (N=70)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Cecal obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Jejunal perforation (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Cardiac troponin T increased (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2)
Speech disorder (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab, Cyclophosphamide) (N=70)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 32 (105)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (3)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (5)
Pericardial effusion (Cardiac disorders) | 1 (16)
Sinus tachycardia (Cardiac disorders) | 4 (6)
Ear pain (Ear and labyrinth disorders) | 2 (3)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 2 (24)
Hearing test abnormal (Ear and labyrinth disorders) | 2 (18)
Tinnitus (Ear and labyrinth disorders) | 5 (58)
Cataract (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 3 (4)
Eye pain (Eye disorders) | 1 (1)
Flashing vision (Eye disorders) | 2 (11)
Vision blurred (Eye disorders) | 5 (8)
Abdominal distension (Gastrointestinal disorders) | 18 (47)
Abdominal pain (Gastrointestinal disorders) | 43 (142)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 37 (129)
Diarrhea (Gastrointestinal disorders) | 27 (99)
Dry mouth (Gastrointestinal disorders) | 4 (16)
Dyspepsia (Gastrointestinal disorders) | 17 (80)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 2 (12)
Esophagitis (Gastrointestinal disorders) | 1 (5)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (12)
Gastritis (Gastrointestinal disorders) | 2 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 7 (31)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 9 (48)
Ileus (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (4)
Mucositis oral (Gastrointestinal disorders) | 16 (38)
Nausea (Gastrointestinal disorders) | 44 (115)
Oral hemorrhage (Gastrointestinal disorders) | 5 (21)
Oral pain (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 4 (13)
Rectal fistula (Gastrointestinal disorders) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (8)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (3)
Tooth disorder (Gastrointestinal disorders) | 7 (26)
Toothache (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 29 (57)
Chest pain (General disorders) | 5 (15)
Chills (General disorders) | 10 (11)
Disease progression (General disorders) | 41 (41)
Edema limbs (General disorders) | 8 (33)
Fatigue (General disorders) | 63 (408)
Fever (General disorders) | 9 (10)
Flu-like symptoms (General disorders) | 5 (6)
General symptom (General disorders) | 4 (5)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 13 (36)
Hypersensitivity (Immune system disorders) | 3 (3)
Bladder infection (Infections and infestations) | 3 (21)
Conjunctivitis infective (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 6 (9)
Infectious colitis (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 5 (8)
Phlebitis infective (Infections and infestations) | 2 (4)
Pneumonia (Infections and infestations) | 3 (7)
Rhinitis infective (Infections and infestations) | 2 (4)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 4 (12)
Vaginal infection (Infections and infestations) | 2 (2)
Vulvitis (Infections and infestations) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 3 (6)
Fracture (Injury, poisoning and procedural complications) | 4 (7)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 14 (41)
Alanine aminotransferase increased (Investigations) | 25 (109)
Alkaline phosphatase increased (Investigations) | 31 (97)
Amylase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 29 (62)
Coagulopathy (Investigations) | 1 (2)
Creatine phosphokinase increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 25 (162)
Haptoglobin decreased (Investigations) | 1 (1)
Hyperbilirubinemia (Investigations) | 3 (6)
Hypercholesterolemia (Investigations) | 1 (1)
INR increased (Investigations) | 5 (6)
Laboratory test abnormal (Investigations) | 1 (1)
Leukopenia (Investigations) | 29 (114)
Lymphopenia (Investigations) | 44 (351)
Neutrophil count decreased (Investigations) | 18 (40)
Platelet count decreased (Investigations) | 10 (65)
Serum cholesterol increased (Investigations) | 1 (2)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 7 (44)
Anorexia (Metabolism and nutrition disorders) | 28 (73)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (19)
Hypercalcemia (Metabolism and nutrition disorders) | 13 (27)
Hyperglycemia (Metabolism and nutrition disorders) | 19 (53)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (16)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 7 (10)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (24)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 13 (27)
Hypomagnesemia (Metabolism and nutrition disorders) | 26 (165)
Hyponatremia (Metabolism and nutrition disorders) | 23 (62)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (8)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (4)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (4)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (74)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (82)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 26 (182)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (73)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (17)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (15)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (27)
Dizziness (Nervous system disorders) | 14 (38)
Extrapyramidal disorder (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 42 (234)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (5)
Neurological disorder NOS (Nervous system disorders) | 1 (2)
Olfactory nerve disorder (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (127)
Sinus pain (Nervous system disorders) | 1 (6)
Speech disorder (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 6 (30)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 22 (124)
Confusion (Psychiatric disorders) | 1 (6)
Depression (Psychiatric disorders) | 13 (62)
Insomnia (Psychiatric disorders) | 19 (145)
Bladder pain (Renal and urinary disorders) | 2 (5)
Cystitis (Renal and urinary disorders) | 2 (5)
Hemoglobinuria (Renal and urinary disorders) | 1 (3)
Hemorrhage urinary tract (Renal and urinary disorders) | 10 (38)
Kidney pain (Renal and urinary disorders) | 2 (31)
Protein urine positive (Renal and urinary disorders) | 2 (13)
Proteinuria (Renal and urinary disorders) | 30 (137)
Ureteric obstruction (Renal and urinary disorders) | 1 (6)
Urethral hemorrhage (Renal and urinary disorders) | 2 (2)
Urethral pain (Renal and urinary disorders) | 2 (14)
Urinary frequency (Renal and urinary disorders) | 5 (9)
Urinary incontinence (Renal and urinary disorders) | 2 (12)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 2 (8)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 2 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (2)
Vaginal pain (Reproductive system and breast disorders) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 18 (57)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (45)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (112)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 11 (23)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 9 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (115)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (23)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (17)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (13)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (12)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (30)
Rash desquamating (Skin and subcutaneous tissue disorders) | 12 (25)
Skin disorder (Skin and subcutaneous tissue disorders) | 6 (20)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 7 (17)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 2 (2)
Hemorrhage (Vascular disorders) | 3 (6)
Hot flashes (Vascular disorders) | 10 (68)
Hypertension (Vascular disorders) | 27 (185)
Hypotension (Vascular disorders) | 1 (1)
Vascular disorder (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less